CLINICAL TRIAL: NCT05123391
Title: Technical Feasibility of a Randomized Pilot Study of Radiosurgery for the Treatment of Non-metastatic Prostate Cancer
Brief Title: Randomized Pilot Study of Radiosurgery for the Treatment of Non-metastatic Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210406002
Record Dates: First submitted 2021-10-27; First posted 2021-11-17 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Prostatic Neoplasms; Radiosurgery; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low-Intermediate favorable risk 5 Fraction SBRT arm (Experimental): 36.25 Gy in 5 fractions to the prostate weekly or every other day
  Interventions: Radiation: External beam image guided radiotherapy
- Low-Intermediate favorable risk 2 Fraction SBRT arm (Experimental): 26 Gy in 2 fractions to the prostate
  Interventions: Radiation: External beam image guided radiotherapy
- Intermediate unfavorable-high risk prostate only SBRT arm (Experimental): 36.25 Gy in 5 fractions to the prostate and seminal vesicles base, weekly or every other day
  Interventions: Radiation: External beam image guided radiotherapy
- Intermediate unfavorable-high risk prostate and pelvis SBRT arm (Experimental): 25 Gy in 5 fractions to the elective pelvic nodes and simultaneous integrated boost to 36.25 Gy in 5 fractions to the prostate and seminal vesicles base, weekly
  Interventions: Radiation: External beam image guided radiotherapy
- Pelvic node positive moderate hypofractionated radiotherapy (Experimental): 44 Gy in 20 daily fractions to the elective pelvic nodes and simultaneous integrated boost to 60 Gy to the prostate and seminal vesicles base and 54 Gy to positive lymph nodes
  Interventions: Radiation: External beam image guided radiotherapy
- Pelvic node positive moderate ultra-hypofractionated radiotherapy (Experimental): 25 Gy in 5 fractions to the elective pelvic nodes and simultaneous integrated boost to 36.25 Gy in 5 fractions to the prostate and seminal vesicles base and to 30 Gy to positive lymph nodes.
  Interventions: Radiation: External beam image guided radiotherapy

INTERVENTIONS:
Radiation: External beam image guided radiotherapy — Volumetric modulated arc therapy (VMAT)-Image-guided radiation therapy (IGRT)

SUMMARY:
This is a prospective, interventional pilot study to evaluate the feasibility of randomizing patients diagnosed with prostate cancer to different treatment schemes according to their risk.

Patients with a diagnosis of prostate adenocarcinoma (confirmed by biopsy), without signs of metastasis outside the pelvis in the staging study and without prior radiotherapy (RT) to the pelvic region will be recruited.

The definition of risk group from the international guide National Comprehensive Cancer Network will be used.

* Low risk
* Favorable intermediate risk
* Unfavorable intermediate risk
* High risk The use of hormonal blocking will be at the discretion of each treating physician.

The radiotherapy simulation will be carried out according to the institutional protocol for the treatment of prostate cancer.

According to the risk group of the patients, the following randomization will be carried out:

* Low / intermediate favorable risk: Patients will be randomized to receive SBRT to prostate 36.25 Gy in 5 fractions, alternate days or weekly, with VMAT (technique and 6 Mega-voltage (MV) X-rays vs to SBRT to prostate 26 Gy in 2 fractions, 1 weekly fraction, with VMAT technique and 6 Mv X-rays. The volumes to be treated, ¨Clinical target volume¨ (CTV) will be defined as the prostate, according to the consensus of the Radiation Therapy Oncology Group (RTOG).
* Intermediate unfavorable risk and high risk: Patients will be randomized to receive SBRT to the prostate and seminal vesicles, 36.25 Gy in 5 fractions, alternate days or weekly, with VMAT technique and 6 MV X-rays vs SBRT to pelvis scheme of 25 Gy in 5 fractions with simultaneous integrated boost up to 36.25 to the prostate and seminal vesicles, with the same technique.
* Patients with positive pelvic node: Will be randomized to moderate hypofractionated RT , completing a dose of 44 Gy in 20 fractions to the pelvis with a simultaneous integrated boost up to 54-60 Gy in 20 fractions to metastatic lymphadenopathy and prostate with seminal vesicles, completing 60 Gy to prostate and seminal vesicles or to ultra hypofractionated RT to the prostate and macroscopic lymphadenopathy to 35 and 30-35 Gy respectively and 25 Gy in 5 fractions to the elective nodal areas.

DETAILED DESCRIPTION:
Background

Prostate cancer is the most common non-cutaneous neoplasm in men both worldwide and in Chile, being the third cause of death in our country. Radiation therapy (RT) is a well-validated curative treatment alternative for prostate cancer, generally being combined with androgen deprivation therapy in intermediate and high risk patients. Dose escalation of RT improves event-free survival and the need for new therapies in the future (continuous androgen deprivation). This dose escalation strategy involves long-term treatments (7 to 8 weeks) with high operational cost for the patient (stays, transportation, etc.) and radiotherapy services.

Hypofractionated RT (reduction of treatment fractions) has shown a similar safety profile and oncological results equivalent to dose escalation in several phase III studies, allowing the total treatment time to be reduced to 4-5 weeks and thus be a more convenient treatment for patients and the radiotherapy department. In the same way, radiosurgery or stereotaxic body radiotherapy (SBRT), is a highly conformed RT technique that significantly reduces the total treatment time (1-2 weeks of treatment). In recent years, the safety and efficacy of SBRT in low- and intermediate-risk prostate cancer has been proven in phase III studies; and in high-risk patients, its low toxicity profile and good biochemical control have been demonstrated in a systematic review. Since this radiotherapy technique has recently been introduced into clinical practice, there are different approaches in relation to the number of fractions used and volumes to be treated.

A pilot study was designed to evaluate the technical feasibility of implementing the randomization of patients who are candidates for radiosurgery between schemes previously used in the literature according to their risk and stage: 2 vs 5 fractions in low / intermediate risk patients include or not pelvic treatment in high-risk patients and a moderate hypofractionated treatment regimen of 20 vs 5 fractions in cN1 or higher patients.

Methods

This is a prospective, interventional pilot study to evaluate the feasibility of randomizing patients diagnosed with prostate cancer to different treatment schemes according to their risk.

Patients with a diagnosis of prostate adenocarcinoma (confirmed by biopsy), without signs of metastasis outside the pelvis in the staging study and without prior RT to the pelvic region will be recruited.

The definition of risk group from the international guide National Comprehensive Cancer Network will be used.

* Low risk
* Favorable intermediate risk
* Unfavorable intermediate risk
* High risk

The use of hormonal blocking will be at the discretion of each treating physician.

The radiotherapy simulation will be carried out according to the institutional protocol for the treatment of prostate cancer.

According to the risk group of the patients, the following randomization will be carried out:

* Low / intermediate favorable risk: Patients will be randomized to receive SBRT to prostate 36.25 Gy in 5 fractions, alternate days or weekly, with Volumetric modulated arc therapy technique (VMAT) and 6 Mv X-rays vs to SBRT to prostate 26 Gy in 2 fractions, 1 weekly fraction, with VMAT technique and 6 Mv X-rays. The volumes to be treated, ¨clinical target volume¨ (CTV) will be defined as the prostate, according to the consensus of the RTOG.
* Intermediate unfavorable risk and high risk: Patients will be randomized to receive SBRT to the prostate and seminal vesicles, 36.25 Gy in 5 fractions, alternate days or weekly, with VMAT technique and 6 Megavolts MV X-rays vs SBRT to pelvis scheme of 25 Gy in 5 fractions with simultaneous integrated boost up to 36.25 to the prostate and seminal vesicles, with the same technique.
* Patients with positive regional pelvic nodes: Patients will be randomized to moderate hypofractionated RT, completing a dose of 44 Gy in 20 fractions to the pelvis with a simultaneous integrated boost up to 54-60 Gy in 20 fractions to metastatic lymphadenopathy and prostate with seminal vesicles, completing 60 Gy to prostate and seminal vesicles or to ultra-hypofractionated RT to the prostate and macroscopic lymphadenopathy to 35 and 30-35 Gy respectively and 25 Gy in 5 fractions to the elective nodal areas.

Contouring of the prostate, seminal vesicles and pelvis will be performed according to the consensus of the NRG Oncology Group.

The treatment will be delivered at the Radiotherapy Service of the Cancer Center, in the a linear accelerator unit with daily verification images.

Before starting treatment and during follow ups urinary symptoms will be assessed by the International Prostate Symptom Score (IPSS) scale, and the The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) and quality of life with "The Expanded Prostate Cancer Index Composite "v2.0 (EPIC 2.0), and the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire-30 (QLQ-30 and QLQ-PR25). The patient will be monitored weekly during the delivery of radiation therapy to assess acute toxicity.

The last day of radiotherapy will be counted as day zero, and the patient will be monitored after 30 days, then every 6 months with IPSS, CTCAE, EPIC, QLQ-30, QLQ-PR25 and prostate specific antigen (PSA) according to the follow-up protocol.

A randomization feasibility trial was designed for each of the 3 groups of patients, assigned 1: 1 for different interventions in each group. The CONSORT recommendations and the Lewis et al method were followed to calculate the sample size and define the feasibility objectives, respectively.

Three key objectives were defined to assess the feasibility of the trial: recruitment acceptance (Percentages of selected patients recruited), treatment fidelity, and patient retention (follow-up). An exact 1-tailed binomial test was used with 5% significance and 80% power.

The feasibility criteria will correspond to:

1. Recruitment: At least 80% (green indicator) of eligible patients must be recruited, the trial will not be feasible if recruitment uptake is less than or equal to 40% (red indicator).
2. Treatment fidelity: A high level of treatment fidelity is required with 80% or more (green indicator) of patients receiving the treatment plan without major protocol deviations, if less than 40% of patients comply with this indicator (red indicator) the test will not be feasible.
3. Follow-up: At least 80% (green indicator) of the patients must remain in follow-up to meet feasibility, if 40% or less (red indicator) comply with retention, the trial will not be feasible.

For this feasibility study a sample size of 30 patients is calculated (5 for each branch of the protocol).

This sample size calculation and feasibility criteria will be used for each of the 3 groups of patients.

In the case an indicator in the red zone the study will stop, in the case all the indicators are in green, a follow up study will be carried out, in the case any indicator is yellow (between 80% and 40%), the pertinent corrections will be made to proceed to a further study.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed prostate cancer
* Disease confined to the pelvis by imaging CT (CT scan of chest, abdomen and pelvis and bone scan or prostate specific membrane antigen positron emission tomography (PET-PSMA) if required according to local guidelines)
* Eastern Cooperative Oncology Group (ECOG) performance 0-1
* Eligible for curative radiotherapy

Exclusion Criteria:

* Metastasis beyond the pelvis
* Poor performance ECOG 2-4
* Cannot follow directions to prepare for simulation (bladder filling and rectal emptying)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 12 months
  Percentage of screened patients eligible recruited
Treatment protocol fidelity | 12 months
  Percentage of recruited patients receiving treatment according to protocol
Follow up | 12 months
  Percentage of recruited patients effectively followed according to protocol

SECONDARY OUTCOMES:
Biochemical control | 24 months
  Failure defined according Phoenix definition (rise by 2 ng/mL or more above the nadir PSA)
Change From Baseline In Quality Of Life (QoL) Total Score As Assessed By The Global Health Domain Of The European Organization Of Research And Treatment Of Cancer (EORTC)-Quality Of Life Questionnaire (QLQ)-C30 | 6,12 and 24 months
  The EORTC QLQ-C30 core measurement was used to capture distal outcomes, including physical, social functioning, and overall health-related quality of life. The questionnaire incorporates 30 questions comprising nine multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 3 symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality of life scale. All raw domain scores are linearly transformed to a 0-100 scale. The global health and quality of life domain is presented. An increase in activity or functioning scores indicates improvement (higher/healthier level of functioning) and a decrease in symptom scores indicates improvement (lower level of symptoms/problems)
Change From Baseline In QoL Total Score As Assessed By The EORTC-QLQ-PR25 Sexual Activity And Functioning And Hormonal-Treatment-Related Symptom Subdomains. | 6, 12 and 24 months
  Subscales for assessment of hormonal treatment-related symptoms (6 items) and sexual activity and function (6 items) from the EORTC-QLQ-PR25 25-item prostate cancer module of the EORTC are presented. Questions used 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale. An increase in activity or functioning scores indicates improvement (higher/healthier level of functioning) and a decrease in symptom scores indicates improvement (lower level of symptoms/problems).

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile